CLINICAL TRIAL: NCT03800615
Title: Iatrogenic Impairment of Urethral Coitus Owing to Midurethral Sling Procedure in a Woman With Vaginal Agenesis.
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 107183-C
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-01

CONDITIONS: Stress Urinary Incontinence; Vaginal Agenesis
MeSH Terms: conditions — Urinary Incontinence, Stress; Vagina, absence of

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cut the sling — Cut the mid-urethral sling for stress urinary incontinence

SUMMARY:
To report a case of impairment urethral coitus after the midurethral sling procedure

DETAILED DESCRIPTION:
To report a case of impairment urethral coitus after the midurethral sling procedure.

ELIGIBILITY:
Inclusion Criteria:

* midurethral sling procedure for stress urinary incontinence
* woman with vaginal agenesis.

Exclusion Criteria:

* Nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A 59-year-old woman had previous history of hysterectomy due to nonfunctional uterine obstruction at 19 years old and urinary incontinence status post transvaginal tape procedure at 45 years old with clinical symptoms of difficulty in urethral coitus after midurethral sling procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sexual function | 1 year
  Asking the patient whether she can resume sexual intercourse or not after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided